CLINICAL TRIAL: NCT03998150
Title: Holmium Laser Enucleation Versus Bipolar Plasmakinetic Enucleation of a Large Volume Benign Prostatic Hyperplasia: a Randomised Controlled Study
Brief Title: Holmium Laser vs Bipolar Enucleation of a Large Volume BPH: a Randomised Controlled Study
Acronym: BPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSheemy, Professor of Urology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 61647
Record Dates: First submitted 2019-06-14; First posted 2019-06-26 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: BPH With Urinary Obstruction; Male
Keywords: BPH; enucleation; Prostate; LUTS; IPSS; quality of life; Large prostate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HoLEP holmium laser enucleation of the prostate (Active Comparator): holmium laser enucleation of the prostate
  Interventions: Procedure: Holmium laser enucleation of the prostate
- BPEP bipolar plasmakinetic enucleation of the prostate (Active Comparator): bipolar plasmakinetic enucleation of the prostate
  Interventions: Procedure: Bipolar plasma kinetic enucleation of the prostate

INTERVENTIONS:
Procedure: Holmium laser enucleation of the prostate — cystoscopic transurethral enucleation of the prostate using Holmium laser (Asclepion MultiPulse HoPlus 110W and Lumenis pulse 100W and 120W)
  Other Names: HoLEP
  Arms: HoLEP holmium laser enucleation of the prostate
Procedure: Bipolar plasma kinetic enucleation of the prostate — cystoscopic transurethral enucleation of the prostate using bipolar plasma kinetic energy (KLS Martin Maxium or Covidien Force Triad)
  Other Names: BPEP
  Arms: BPEP bipolar plasmakinetic enucleation of the prostate

SUMMARY:
To compare bipolar plasmakinetic enucleation versus holmium laser enucleation for management of large BPH.

DETAILED DESCRIPTION:
To compare safety and efficacy of bipolar plasmakinetic enucleation (BPEP) versus holmium laser enucleation (HoLEP) for management of large BPH (>80gm).

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from LUTS secondary to infravesical obstruction from BPH
* failed medical treatment
* International Prostate Symptom Score (IPSS) > 13
* a peak urinary flow rate (Qmax) < 15 ml/sec
* a prostate size ≥ 80 gm

Exclusion Criteria:

* presence of a urethral stricture
* neurological disorder
* bladder cancer
* prostate cancer
* previous history of bladder neck surgery or TURP

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
hemoglobin drop postoperatively (gm/dL) | Immediate postoperatively
  difference in hemoglobin concentration postoperatively vs preoperatively
operative time | during surgery
  operative time in minutes

SECONDARY OUTCOMES:
complications (%) | one year
  intraoperative and postoperative complications including blood transfusion, capsular perforation, irritative symptoms, SUI, urethral stricture, bladder neck contracture, urinary retention.
urine flow | one year
  Qmax (ml/s),
post-voiding residual urine | one year
  postvoiding residual urine (ml)
International prostate symptom score (IPSS) | one year
  an international commonly used score ranging from 0 - 35 (the worst is 35) evaluating voiding and storage urinary symptoms using 7 questions each one is scored from 0 to 5 according to severity of symptom
Quality of life (QoL) section of International prostate symptom score (IPSS) | one year
  one question scored from 0 up to 6 (6 is worst)

CONTACTS AND LOCATIONS:
Overall Officials: enmar I Habib, Prof., Study Director — Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Habib E, Ayman LM, ElSheemy MS, El-Feel AS, Elkhouly A, Nour HH, Badawy MH, Elbaz AG, Roshdy MA. Holmium Laser Enucleation vs Bipolar Plasmakinetic Enucleation of a Large Volume Benign Prostatic Hyperplasia: A Randomized Controlled Trial. J Endourol. 2020 Mar;34(3):330-338. doi: 10.1089/end.2019.0707. Epub 2020 Feb 28. PMID 31813283